CLINICAL TRIAL: NCT07173725
Title: Octenidine Versus Chlorhexidine as the Final Irrigant in Single-visit Endodontics: a Randomized Clinical Trial of Early Postoperative Pain
Brief Title: The Effect of Using Octenidine Hydrochloride as a Final Irrigation Solution on Teeth With Asymptomatic Apical Periodontitis on Postoperative Pain and Treatment Success: A Prospective Randomized Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08.03.2023-E.99606
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Apical Periodontitis; Postoperative Pain
Keywords: Endodontics; Root canal treatment; Final irrigant; Single-visit endodontics; Chlorhexidine; Octenidine
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative | interventions — octenidine; Solutions; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group, single-centre endodontic trial; single-visit treatment; final irrigant: octenidine vs chlorhexidine.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Irrigants prepared by a third party in identical opaque A/B syringes; allocation concealed with SNOSE; participants, care provider (operator), and outcomes assessor were blinded; A/B code broken only after database lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Octenidine 0.1% final irrigant (Experimental): Single-visit root canal treatment with octenidine dihydrochloride 0.1% as the final irrigant. The irrigant was sonically activated using three 20-second cycles; the solution was refreshed with 2 mL between cycles (approximate total 6 mL). Delivery through a side-vented needle positioned short of the working length. The final irrigant was administered once, during the final irrigation phase. All other procedural steps were identical to the comparator arm.
  Interventions: Drug: Octenidine dihydrochloride 0.1%
- Chlorhexidine 2% final irrigant (Active Comparator): Single-visit root canal treatment with chlorhexidine 2% as the final irrigant. The irrigant was sonically activated using the same protocol as the experimental arm: three 20-second cycles with the solution refreshed with 2 mL between cycles (approximate total 6 mL). Delivery through a side-vented needle positioned short of the working length. The final irrigant was administered once, during the final irrigation phase. All other procedural steps were identical to the experimental arm.
  Interventions: Drug: Chlorhexidine 2%

INTERVENTIONS:
Drug: Octenidine dihydrochloride 0.1% — Final intracanal irrigant (aqueous solution); single administration during the final irrigation phase. Sonic activation performed in three 20-second cycles; solution refreshed with 2 mL between cycles (approximate total 6 mL per canal). Delivered through a side-vented needle positioned short of the working length.
  Other Names: OCT; Octenidine 0.1% solution
  Arms: Octenidine 0.1% final irrigant
Drug: Chlorhexidine 2% — Final intracanal irrigant (aqueous solution); single administration during the final irrigation phase. Sonic activation performed in three 20-second cycles; solution refreshed with 2 mL between cycles (approximate total 6 mL per canal). Delivered through a side-vented needle positioned short of the working length.
  Other Names: CHX; Chlorhexidine 2% solution
  Arms: Chlorhexidine 2% final irrigant

SUMMARY:
This single-centre, randomized, parallel-group clinical trial compared two commonly used final irrigants in single-visit root canal treatment: octenidine dihydrochloride (OCT) and chlorhexidine (CHX). Adults with single-rooted, single-canal teeth diagnosed with asymptomatic apical periodontitis were treated in one visit under local anaesthesia and rubber-dam isolation. After shaping with sodium hypochlorite and smear-layer removal with EDTA, the assigned final irrigant was delivered and sonically activated. In both groups, OCT 0.1 percent or CHX 2 percent was activated using three 20-second cycles, and the solution was refreshed with 2 mL between cycles (approximate total 6 mL). Postoperative pain was recorded by participants on an 11-point Numeric Rating Scale (0 = no pain, 10 = worst pain) at 6, 12, 24, and 48 hours. The primary outcome was pain at 48 hours. Secondary outcomes were pain at earlier time points, use of rescue analgesics within 0-48 hours, and unplanned urgent care within 48 hours. The aim was to determine whether OCT reduces early postoperative pain compared with CHX when used as the final irrigant in single-visit endodontics.

DETAILED DESCRIPTION:
Design and setting. Prospective, randomized, parallel-group, blinded clinical trial conducted at a university dental hospital (Istanbul, Turkey). All treatments were completed in a single visit by an experienced endodontist using local anaesthesia and rubber-dam isolation.

Participants. Adults (18 years or older) with single-rooted, single-canal teeth diagnosed with asymptomatic apical periodontitis on periapical radiographs were eligible. Exclusion criteria included symptomatic apical periodontitis or acute abscess, previous root-canal treatment of the study tooth, systemic conditions interfering with pain assessment or requiring antibiotic prophylaxis, pregnancy or lactation, known allergy to study materials, and use of analgesics or anti-inflammatory drugs within 12 hours before treatment. One patient contributed one tooth.

Randomization, allocation concealment, and masking. Participants were randomized 1:1 to OCT or CHX using computer-generated permuted blocks with stratification by baseline pain (NRS <= 3 vs > 3). Allocation was concealed with sequentially numbered, opaque, sealed envelopes. Irrigants were prepared by a third party in identical opaque syringes labelled A/B. Participants, the care provider (operator), and the outcomes assessor were blinded until database lock.

Interventions. Working length was established with an electronic apex locator and confirmed radiographically when needed. Root canals were prepared with nickel-titanium rotary instruments to size 40/0.04. During shaping, 5.25 percent sodium hypochlorite was used (approximately 2 mL after each instrument change). The smear layer was removed with 17 percent EDTA (about 10 mL) activated with a sonic device, followed by saline. For the final irrigation, the allocated solution was delivered and sonically activated using the same protocol in both groups: OCT 0.1 percent or CHX 2 percent, activated in three 20-second cycles with the solution refreshed with 2 mL between cycles (approximate total 6 mL). A side-vented needle was placed short of the working length. Root-canal obturation was completed in the same session using gutta-percha and an epoxy resin-based sealer with cold lateral compaction. Access cavities were restored with a resin composite. Rescue analgesics were permitted as needed and recorded by patients.

Outcomes. Primary outcome: patient-reported pain on the 0-10 NRS at 48 hours after treatment. Secondary outcomes: NRS pain at 6, 12, and 24 hours; total rescue analgesic consumption from 0 to 48 hours; and unplanned urgent care or adverse events within 48 hours.

Sample size and analysis plan. The a priori sample-size calculation assumed a between-group difference of 1.0 NRS unit (SD 2.0), alpha 0.05, and power 0.80, yielding 100 participants; allowing for attrition, the target was 120. Analyses compared groups at 48 hours and evaluated pain trajectories over time using mixed-effects methods with fixed effects for group and time and a random intercept for participant. Two-sided p < 0.05 was considered statistically significant.

Oversight. The protocol was approved by the Bezmialem Vakif University Clinical Research Ethics Committee (approval E.99606). The trial was conducted in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years (inclusive)
* Single-rooted, single-canal tooth
* Diagnosis of asymptomatic apical periodontitis on periapical radiographs
* Able and willing to provide written informed consent
* Able to complete a 48-hour pain diary (6 h, 12 h, 24 h, 48 h)

Exclusion Criteria:

* Symptomatic apical periodontitis or acute apical abscess
* Previous root canal treatment of the study tooth
* Systemic condition requiring antibiotic prophylaxis or that interferes with pain assessment
* Pregnancy or lactation
* Known allergy or contraindication to study irrigants/materials
* Use of analgesics or anti-inflammatory drugs within 12 hours before treatment
* Inability to comply with study procedures
* More than one eligible tooth (one patient = one tooth rule; a pre-specified index tooth is selected)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Pain at 48 hours (NRS 0-10) | 48 hours after treatment
  Patient-reported pain on the 11-point Numeric Rating Scale (NRS, 0 = no pain, 10 = worst pain). Higher scores indicate worse pain. Assessed using a patient diary. Analysis compares OCT vs CHX at 48 hours; analysis population includes all randomized participants with an available 48 h NRS value.

SECONDARY OUTCOMES:
Pain at 6 hours (NRS 0-10) | 6 hours after treatment
  Patient-reported NRS pain score (0 = no pain, 10 = worst pain). Higher scores indicate worse pain. Assessed using a patient diary; between-group comparison at 6 hours.
Pain at 12 hours (NRS 0-10) | 12 hours after treatment
  Patient-reported NRS pain score (0 = no pain, 10 = worst pain). Higher scores indicate worse pain. Assessed using a patient diary; between-group comparison at 12 hours.
Pain at 24 hours (NRS 0-10) | 24 hours after treatment
  Patient-reported NRS pain score (0 = no pain, 10 = worst pain). Higher scores indicate worse pain. Assessed using a patient diary; between-group comparison at 24 hours.
Rescue analgesic consumption (0-48 hours) | 0 to 48 hours after treatment
  Number of self-reported rescue analgesic doses taken from 0 to 48 hours after treatment (any medication allowed per routine care). Participants recorded type, dose, and timing in a diary. Higher counts indicate greater analgesic use.
Unplanned urgent care within 48 hours | Up to 48 hours after treatment
  Count of participants who required unplanned urgent dental care (eg, unscheduled clinic visit or phone consultation requiring prescription) within 48 hours after treatment. Reported as number and proportion of participants.
Adverse events within 48 hours (postoperative flare-up and other events) | Up to 48 hours after treatment
  Occurrence of any adverse event within 48 hours after treatment, including postoperative flare-up requiring unplanned care. Reported as number and proportion of participants with at least one event; serious and non-serious events summarized separately.

OTHER OUTCOMES:
Analgesic-free participants (0-48 hours) | 0 to 48 hours after treatment
  Proportion of participants who took no rescue analgesics from 0 to 48 hours after treatment (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: fatma B peker, dds, Principal Investigator — Department of Endodontics, Bezmialem Vakif University, Istanbul, Turkey
Locations (1):
- Bezmialem Vakif University Dental Hospital - Department of Endodontics, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Bezmialem Vakif University - study site — http://bezmialem.edu.tr/